CLINICAL TRIAL: NCT00529594
Title: Analgesic Effect of Etoricoxib (ARCOXIA®) 120MG During Retinal Laser Photocoagulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 519/06
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Last update posted 2007-09-14 (Estimated); Status verified 2007-03

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Laser Photocoagulation; Pain relief
MeSH Terms: interventions — Control Groups; Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Placebo Comparator): Patients who received placebo
  Interventions: Drug: placebo (Control Group)
- Treatment Group (Active Comparator): Patients who received etoricoxib 120 mg
  Interventions: Drug: Etoricoxib (Treatment Group)

INTERVENTIONS:
Drug: placebo (Control Group) — Both medication have been given to the patients in both groups 1 hour prior the laser photocoagulation
  Arms: Control Group
Drug: Etoricoxib (Treatment Group) — Both medication have been given to the patients in both groups 1 hour prior the laser photocoagulation
  Other Names: Etoricoxib 120mg is Arcoxia 120mg
  Arms: Treatment Group

SUMMARY:
The study wants to show if the medication etoricoxib 120 mg have reduces the patients pain during the laser photocoagulation, for diabetic retinopathy.

DETAILED DESCRIPTION:
To do so we compare two group of patients, randomized 1:1, one use the medication(etoricoxib) and other use placebo and they quantify the pain using the Pain visual analogue scale

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetic retinopathy that needs laser photocoagulation for the first time

Exclusion Criteria:

* Younger than 17
* Signs and symptoms of liver dysfunction or abnormal liver function tests
* Gastrointestinal diseases
* Pregnant women
* Edema
* Pre-existing cardiac insufficiency

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-08; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The group taking the etoricoxib feel less pain then the group taking placebo | After each laser session

CONTACTS AND LOCATIONS:
Overall Officials: Vinicius P Nascimento, MD, Principal Investigator — Clinica Oftalmologica do Hospital das Clinicas da Universidade de São Paulo
Locations (1):
- Clinica Oftalmologica do Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, São Paulo, Brazil